CLINICAL TRIAL: NCT01558674
Title: A Two Part, Open-label, Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MK-7145 in Patients With Renal Insufficiency (Part I) and Heart Failure With Renal Insufficiency (Part II)
Brief Title: A Study of MK-7145 in Participants With Renal Insufficiency (Part I) and Heart Failure With Renal Insufficiency (Part II) (MK-7145-011)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7145-011
Record Dates: First submitted 2012-03-16; First posted 2012-03-20 (Estimated); Results first posted 2017-03-03 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-08

CONDITIONS: Renal Impairment; Heart Failure
MeSH Terms: conditions — Renal Insufficiency; Heart Failure | interventions — MK-7145; Furosemide; Torsemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- MK-7145 8 mg (Part I:Period 1) (Experimental): Single daily dose of 8 mg MK-7145 for 5 days, capsules, orally administered in a fasted state
  Interventions: Drug: MK-7145
- Furosemide 40 mg (Part I:Period 2) (Active Comparator): Two daily doses of one 40 mg Furosemide tablet for 5 days administered in a fasted state
  Interventions: Drug: Furosemide
- MK-7145 16 mg (Part I:Period 3) (Experimental): Single daily dose of 16 mg MK-7145 for 5 days, capsules, orally administered in a fasted state
  Interventions: Drug: MK-7145
- Furosemide/Torsemide Run-in (Part II:Period1) (Active Comparator): Run-in of stable, clinically optimized maintenance dose regimen of furosemide or torsemide for at least 2 weeks
  Interventions: Drug: Furosemide; Drug: Torsemide
- MK-7145 10 mg (Part II:Period 2) (Experimental): Single daily dose of 10 mg MK-7145 for 14 days, capsules, orally administered in a fasted state
  Interventions: Drug: MK-7145
- MK-7145 16 mg (Part II:Period 3) (Experimental): Single daily dose of 16 mg MK-7145 for 14 days, capsules, orally administered in a fasted state
  Interventions: Drug: MK-7145
- MK-7145 24 mg (Part II:Period 4) (Experimental): Single dose of 24 mg MK-7145 for 28 days, capsules, orally administered in a fasted state
  Interventions: Drug: MK-7145

INTERVENTIONS:
Drug: MK-7145
  Arms: MK-7145 10 mg (Part II:Period 2); MK-7145 16 mg (Part I:Period 3); MK-7145 16 mg (Part II:Period 3); MK-7145 24 mg (Part II:Period 4); MK-7145 8 mg (Part I:Period 1)
Drug: Furosemide
  Other Names: Lasix
  Arms: Furosemide 40 mg (Part I:Period 2); Furosemide/Torsemide Run-in (Part II:Period1)
Drug: Torsemide
  Arms: Furosemide/Torsemide Run-in (Part II:Period1)

SUMMARY:
Part I is a 3-period, active comparator-controlled, fixed sequence study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of MK-7145 compared to furosemide in participants with moderate-to-severe renal insufficiency (RI) without heart failure (HF). Primary hypothesis for Part I is that at least one well-tolerated dose of MK-7145 will produce a greater 24hr urinary excretion of sodium (UNa) on the 1st day of MK-7145 dosing than 80 mg furosemide (on the 1st day of furosemide dosing) in participants with moderate-to-severe RI. If MK-7145 is safe at natriuretic doses in RI in Part I of this study, MK-7145 will be investigated in participants with heart failure (HF) and RI (Part II).

Part II is 4 period, fixed sequence, active comparator controlled (in Period 1), titration (in Periods 2, 3 and 4) study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of a titration regimen of MK-7145 compared to an optimized stable maintenance regimen of furosemide or torsemide in participants with New York Heart Association (NYHA) Class II and III heart failure and moderate or severe renal insufficiency. The primary hypothesis for Part II is that at least one dose of MK-7145, titrated according to a fixed dose titration regimen, will be associated with a reduction in N-terminal pro-brain natriuretic peptide (NT-proBNP) compared to furosemide or torsemide (at 24 hours post morning dose on the last dosing day of each period) in participants with NYHA class II/III HF with moderate or severe RI.

ELIGIBILITY:
Inclusion Criteria:

Parts I and II

* If female, must be of non-child bearing potential or, if of child-bearing potential agrees to use at least 2 acceptable contraceptive measures
* Body Mass Index (BMI) >=17.5 and <=38 kg/m^2
* No present history of clinically significant uncontrolled arrhythmias on electrocardiogram (ECG)
* Nonsmoker or a light smoker consuming up to an average of 20 cigarettes (or equivalent tobacco product) per day.

Part I Only

- Estimated creatinine clearance of ≤45 mL/min.

Part II Only

* Class II or III heart failure as specified by the New York Heart Association (NYHA) functional classification for heart failure with NT-proBNP >=1000 pg/mL on clinically optimized therapy with a stable dose (for at least 2 weeks) of furosemide or torsemide
* Estimated creatinine clearance of ≤45 mL/min

Exclusion Criteria:

Parts I and II

* Mentally or legally institutionalized and/or incapacitated, has significant emotional problems or has a history of a clinically significant psychiatric disorder over the last 5 years. This includes any mood disorder requiring concomitant use of lithium
* Diagnosed with acute coronary syndrome or acute cardiovascular (CV) event, or has been hospitalized for HF exacerbation within less than 3 months of study entry
* Unstable angina pectoris
* Diabetes requiring high dose peroxisome proliferator-activated receptor (PPAR) antagonist (e.g. >30 mg of pioglitazone) or unstable insulin use
* Infectious disease requiring concomitant use of aminoglycosides
* Low plasma potassium (hypokalemia)
* Recent (within 6 months) history of stroke, uncontrolled seizures, or uncontrolled major neurological disorder
* Urinary retention, hydronephrosis or hydroureter
* Active nephrocalcinosis, nephrolithiasis, or hypercalciuria
* Functional disability that can interfere with rising from a semi-recumbent position to the standing position
* History of malignant neoplastic disease
* Unable to refrain from the use of medication, including prescription and non-prescription drugs such as high-dose aspirin (≥325 mg/day), non-steroidal anti-inflammatory drugs (NSAIDs), human immunodeficiency virus (HIV) protease inhibitors (ritonavir, indinavir, nelfinavir), macrolide antibiotics (erythromycin, telithromycin, clarithromycin), chloramphenicol, azole antifungals (fluconazole, ketoconazole, itraconazole, nefazodone, aprepitant, verapamil, diltiazem, etc.), anticonvulsants and mood stabilizers (e.g., phenytoin, carbamazepine, oxcarbazepine), barbiturates (phenobarbital), HIV non-nucleoside reverse transcriptase inhibitors (efavirenz, nevirapine, etravirine), rifampicin, modafinil, St John's wort, cyproterone (antiandrogen, progestin), etc. beginning approximately 2 weeks (or 5 half-lives), prior to administration of the initial dose of study drug, throughout the study (including washout intervals between treatment periods) until the poststudy visit
* Consumes excessive amounts of alcohol, defined as greater than 5 glasses of alcoholic beverages (1 glass is approximately equivalent to: beer [284 mL/10 ounces], wine [125 mL/4 ounces], or distilled spirits [25 mL/1 ounce]) per day
* Consumes excessive amounts, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, or other caffeinated beverages per day
* Had major surgery, donated or lost 1 unit of blood (approximately 500 mL) or participated in another investigational study within 4 weeks
* Regular user of any illicit drugs or has a history of drug (including alcohol) abuse within approximately 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-05-23 (Actual); Primary Completion 2014-12-17 (Actual); Study Completion 2014-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study was terminated early due to lack of efficacy of MK-7145. Only 11 participants were enrolled and dosed in Part 1. Period 3 of Part 1 was not conducted. No participants were enrolled in the planned Part 2 of the study.
Groups:
- MK-7145 8 mg→Furosemide 40 mg 2 x Day (BID)→ MK-7145 16 mg: Part 1: Participants receive 8 mg MK-7145 once daily (QD) for 5 days, then furosemide 40 mg BID for 5 days and then 16 mg MK-7145 QD for 5 days. Each treatment period was separated by a 3-day wash-out.
- Furosemide/Torsemide→MK-7145 10 mg→MK-7145 16 mg→MK-7145 24 mg: Part 2: Participants receive Furosemide/Torsemide for 2 weeks , then 10 mg MK-7145 for 14 days, then MK-7145 16 mg for 14 days and then MK-7145 24 mg for 28 days. Each treatment period was separated by a 3-day wash-out.
Period: Part 1
Arm/Group | MK-7145 8 mg→Furosemide 40 mg 2 x Day (BID)→ MK-7145 16 mg | Furosemide/Torsemide→MK-7145 10 mg→MK-7145 16 mg→MK-7145 24 mg
Started | 11 | 0
Completed | 0 | 0
Not Completed | 11 | 0
Not completed — Study Terminated by Sponsor | 10 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Part 2
Arm/Group | MK-7145 8 mg→Furosemide 40 mg 2 x Day (BID)→ MK-7145 16 mg | Furosemide/Torsemide→MK-7145 10 mg→MK-7145 16 mg→MK-7145 24 mg
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-7145 8 mg→Furosemide 40 mg 2 x Day (BID)→ MK-7145 16 mg | Furosemide/Torsemide→MK-7145 10 mg→MK-7145 16 mg→MK-7145 24 mg | Total
Number analyzed (Participants) | 11 | 0 | 11
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.4 (16.0) |  | 61.4 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 |  | 3
  Male | 8 |  | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in First 24hr Urinary Sodium (UNa) (Part 1)
Description: Urine was collected at Treatment Day -1 and Treatment Day 1 at 0-2, 2-4, 4-6, 6-8, 8-12, 12-24 hour. The 24-hour cumulative natriuresis will be estimated by the amount of sodium excreted into urine over 24 hour period postdose, where amount of sodium is the product of sodium concentration and the volume of urine. The change from baseline in UNa from baseline (Treatment Day -1) and 24 hours post-dose on Treatment Day 1 were calculated.
Time Frame: Baseline (Day -1) and 0-24 hours postdose on Treatment Day 1 of each treatment period
Population: All participants who received at least 1 dose of study drug and who complied with the protocol sufficiently. One participant did not participate for several time intervals on Period 2: Day 8 due to being unwell, and data from this day of this participant were excluded from the analysis. Part 1: Period 3 was not conducted.
Measure: Least Squares Mean (95% Confidence Interval); unit: mEq
Groups:
- MK-7145 8 mg (Part 1: Period 1): 8 mg MK-7145 QD for 5 days, capsules, orally administered in a fasted state
- Furosemide 40 mg BID (Part 1: Period 2): 40 mg Furosemide tablet BID for 5 days administered in a fasted state
- MK-7145 16 mg (Part 1: Period 3): 16 mg MK-7145 QD for 5 days, capsules, orally administered in a fasted state
Arm/Group | MK-7145 8 mg (Part 1: Period 1) | Furosemide 40 mg BID (Part 1: Period 2) | MK-7145 16 mg (Part 1: Period 3)
Number analyzed (Participants) | 11 | 10 | 0
mEq | 11.0 [-18.6 to 40.6] | 109.5 [82.0 to 137.1] |
Statistical Analysis 1: Comparison: MK-7145 8 mg (Part 1: Period 1) vs Furosemide 40 mg BID (Part 1: Period 2); Test type: Superiority or Other; Linear mixed effect model; Difference in Least Squares (LS) Means = -98.5, 95% CI 2-sided [-138.0 to -59.1] — 8-mg MK-7145 LS Mean minus Furosemide LS Mean

2. Primary Outcome: N-terminal Pro B-type Natriuretic Peptide (NT-proBNP) Values at 24 Hours Post Last Morning Dose of Each Period (Part 2)
Description: B-type natriuretic peptide (BNP) is a substance secreted from the ventricles or lower chambers of the heart in response to changes in pressure that occur when heart failure develops and worsens. The level of BNP in the blood increases when heart failure symptoms worsen, and decreases when the heart failure condition is stable. The BNP level in a person with heart failure is higher than in a person with normal heart function. Levels of BNP levels were assessed 24 hours post last morning dose of study drug for each treatment period.
Time Frame: Day 15 for Periods 1, 2, and 3; Day 29 for Period 4
Population: Part 2 of the study was not conducted. No participants were enrolled.
Groups:
- Furosemide/Torsemide (Part 2; Period 1): Stable, clinically optimized maintenance dose regimen of furosemide or torsemide for at least 2 weeks.
- MK-7145 10 mg (Part 2: Period 2): 10 mg of MK-7145 once daily for 14 days
- MK-7145 16 mg (Part 2: Period 3): 14 mg of MK-7145 once daily for 14 days
- MK-7145 24 mg (Part 2: Period 4): 24 mg of MK-7145 once daily for 28 days
Arm/Group | Furosemide/Torsemide (Part 2; Period 1) | MK-7145 10 mg (Part 2: Period 2) | MK-7145 16 mg (Part 2: Period 3) | MK-7145 24 mg (Part 2: Period 4)
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Fold Change From Baseline for Serum Creatinine at 24-hours Post Treatment Day 5 Morning Dose (Part 1)
Description: Blood was collected predose on Treatment Day 1 and at 24 hours post morning dose on Treatment Day 5 to determine serum creatinine levels. Creatinine levels were log transformed and then fold change from baseline was calculated.
Time Frame: Baseline (predose Treatment Day 1) and 24 hours post morning dose on Treatment Day 5 of each treatment period (Part I)
Population: All participants who received at least 1 dose of study drug , who complied with the protocol sufficiently and had data available for endpoint. Part 1: Period 3 was not conducted.
Measure: Geometric Mean (95% Confidence Interval); unit: mg/dL
Groups:
- MK-7145 16 mg (Part I:Period 3): 16 mg MK-7145 QD for 5 days, capsules, orally administered in a fasted state
Arm/Group | MK-7145 8 mg (Part 1: Period 1) | Furosemide 40 mg BID (Part 1: Period 2) | MK-7145 16 mg (Part I:Period 3)
Number analyzed (Participants) | 11 | 10 | 0
mg/dL | 1.30 [1.16 to 1.46] | 1.18 [1.10 to 1.27] |
Statistical Analysis 1: Comparison: MK-7145 8 mg (Part 1: Period 1) vs Furosemide 40 mg BID (Part 1: Period 2); Test type: Superiority or Other; Mixed Linear Effects Model; Geometric Mean Ratio (GMR) = 1.10, 90% CI 2-sided [0.99 to 1.22] — GMR = Geometric mean (GM) MK-7145 8 mg divided by GM Furosemide

4. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to 24 Hours After Dosing (AUC0-24hr) of MK-7145 (Treatment Days 1 and 5: Part 1)
Description: Blood samples for pharmacokinetic analysis were collected on Day 4 (Treatment Day 1) through Day 8 (Treatment Day 5) at the following time points: Predose, 3, 5, 6, 8, 10, 12, 14, 18, 24 , 96, 101, 104, 106, 108, 110 and 120 hours (relative to Day 4 dosing). The AUC0-24 was calculated for Days 1 and 5
Time Frame: up to 24 hours post-dose on Treatment Day 1 and Treatment Day 5
Population: All participants who received at least 1 dose of MK-7145, who complied with the protocol sufficiently and had data available for endpoint. Part 1: Period 3 was not conducted
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*hr
Arm/Group | MK-7145 8 mg (Part 1: Period 1) | MK-7145 16 mg (Part I:Period 3)
Number analyzed (Participants) | 11 | 0
nM*hr
  Treatment Day 1 | 158 (49.2) |
  Treatment Day 5 | 485 (50.4) |

5. Secondary Outcome: Maximum Plasma Concentration (Cmax) of MK-7145 (Treatment Days 1 and 5: Part 1)
Description: Blood samples for pharmacokinetic analysis were collected on Treatment Day 1 through Treatment Day 5 at the following time points: Predose, 3, 5, 6, 8, 10, 12, 14, 18, 24, 96, 101, 104, 106, 108, 110 and 120 hours (relative to Treatment Day 1 dosing). The Cmax was calculated for Treatment Days 1 and 5.
Time Frame: Treatment Day 1 and Treatment Day 5
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | MK-7145 8 mg (Part 1: Period 1) | MK-7145 16 mg (Part I:Period 3)
Number analyzed (Participants) | 11 | 0
nM
  Treatment Day 1 | 10.2 (57.9) |
  Treatment Day 5 | 26.0 (50.3) |

6. Secondary Outcome: Trough Plasma Concentration (Ctrough) of MK-7145 (Treatment Days 1 and 5: Part 1)
Description: Blood samples for pharmacokinetic analysis were collected on Treatment Day 1 through Treatment Day 5 at the following time points: Predose, 3, 5, 6, 8, 10, 12, 14, 18, 24 , 96 , 101, 104, 106, 108, 110 and 120 hours (relative to Treatment Day 1 dosing). The Ctrough for was calculated for Treatment Days 1 and 5
Time Frame: Treatment Day 1 and Treatment Day 5
Population: All participants who received at least 1 dose of MK-7145, who complied with the protocol sufficiently and had data available for endpoint. Ctrough for MK-7145 8 mg arm could not be estimated due to insufficient terminal phase sample. Part 1: Period 3 was not conducted.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | MK-7145 8 mg (Part 1: Period 1) | MK-7145 16 mg (Part I:Period 3)
Number analyzed (Participants) | 11 | 0
nM
  Treatment Day 1 | NA (NA) — Ctrough estimates not available due to lack of data at terminal phase. |
  Treatment Day 5 | NA (NA) — Ctrough estimates not available due to lack of data at terminal phase. |

7. Secondary Outcome: Time to Cmax (Tmax) of MK-7145(Treatment Days 1 and 5: Part 1)
Description: Blood samples for pharmacokinetic analysis were collected on Treatment Day 1 through Treatment Day 5 at the following time points: Predose, 3, 5, 6, 8, 10, 12, 14, 18, 24, 96 , 101, 104, 106, 108, 110 and 120 hours (relative to Treatment Day 1 dosing). The time to Cmax (Tmax) calculated for Treatment Days 1 and 5
Time Frame: Treatment Day 1 and Treatment Day 5
Population: All participants who received at least 1 dose of MK-7145 who complied with the protocol sufficiently and had data available for endpoint. Part 1: Period 3 was not conducted.
Measure: Median (Full Range); unit: hours
Arm/Group | MK-7145 8 mg (Part 1: Period 1) | MK-7145 16 mg (Part I:Period 3)
Number analyzed (Participants) | 11 | 0
hours
  Treatment Day 1 | 10.0 [5.0 to 12.0] |
  Treatment Day 5 | 5.0 [5.0 to 12.0] |

8. Secondary Outcome: Apparent Terminal Half-life (t1/2) of MK-7145 (Part 1)
Description: Blood samples for pharmacokinetic analysis were collected on Treatment Day 1 through Treatment Day 5 at the following time points: Predose, 3, 5, 6, 8, 10, 12, 14, 18, 24, 96, 101, 104, 106, 108, 110 and 120 hours (relative to Treatment Day 1 dosing). The t1/2 was calculated.
Time Frame: Treatment Day 1 and Treatment Day 5
Population: All participants who received at least 1 dose of MK-7145 and who complied with the protocol sufficiently and had data available for endpoint. t1/2 could not be estimated due to insufficient terminal phase sample. Part 1: Period 3 was not conducted.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | MK-7145 8 mg (Part 1: Period 1) | MK-7145 16 mg (Part I:Period 3)
Number analyzed (Participants) | 11 | 0
hours
  Treatment Day 1 | NA [NA to NA] — t1/2 estimates not available due to lack of data at terminal phase. |
  Treatment Day 5 | NA [NA to NA] — t1/2 estimates not available due to lack of data at terminal phase. |

9. Secondary Outcome: Serum Creatinine Measured at 24 Hours Post Last Morning Dose of Each Period (Part 2)
Description: Blood samples were collected at 24 hours post last morning dose of each period to determine serum creatinine levels
Time Frame: Day 15 for Periods 1, 2, and 3; Day 29 for Period 4
Population: No participants were enrolled in Part 2 of the study.
Groups:
- MK-7145 10 mg (Part 2:Period 2): 10 mg of MK-7145 once daily for 14 days
Arm/Group | Furosemide/Torsemide (Part 2; Period 1) | MK-7145 10 mg (Part 2:Period 2) | MK-7145 16 mg (Part 2: Period 3) | MK-7145 24 mg (Part 2: Period 4)
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to 24 Hours After Dosing (AUC0-24hr) of MK-7145 (Part 2)
Description: Blood samples taken at predose, 0.5, 1, 2, 5, 8, 12, 14 and 24 hours postdose on Days 1 and 14 of Period 2 and Day 14 of Periods 3-4 to determine the AUC0-24hr
Time Frame: up to 24 hours post morning dose on Days 1 and 14 of Period 2 and Day 14 of Periods 3 and 4
Population: No participants were enrolled in Part 2 of the study.
Arm/Group | MK-7145 10 mg (Part 2: Period 2) | MK-7145 16 mg (Part 2: Period 3) | MK-7145 24 mg (Part 2: Period 4)
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Maximum Plasma Concentration (Cmax) of MK-7145 (Part 2)
Description: Blood samples taken at predose, 0.5, 1, 2, 5, 8, 12, 14 and 24 hours postdose on Days 1 and 14 of Period 2 and Day 14 of Periods 2-4 to determine the Cmax.
Time Frame: up to 24 hours post morning dose on up to 24 hours post morning dose on Days 1 and 14 of Period 2 and Day 14 of Periods 3 and 4
Population: No participants were enrolled in Part 2 of the study.
Arm/Group | MK-7145 10 mg (Part 2: Period 2) | MK-7145 16 mg (Part 2: Period 3) | MK-7145 24 mg (Part 2: Period 4)
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Trough Plasma Concentration (Ctrough) of MK-7145 (Part 2)
Description: Blood samples taken at predose, 0.5, 1, 2, 5, 8, 12, 14 and 24 hours postdose on Days 1 and 14 of Period 2 and Day 14 of Periods 3 and 4 to determine the Ctrough.
Time Frame: up to 24 hours post morning dose on Days 1 and 14 of Period 2 and Day 14 of Periods 3 and 4
Population: No participants were enrolled in Part 2 of the study.
Groups:
- MK-7145 16 mg: 14 mg of MK-7145 once daily for 14 days
Arm/Group | MK-7145 10 mg (Part 2: Period 2) | MK-7145 16 mg | MK-7145 24 mg (Part 2: Period 4)
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Time to Cmax (Tmax) of MK-7145(Part 2)
Description: Blood samples taken at predose, 0.5, 1, 2, 5, 8, 12, 14 and 24 hours postdose on Days 1 and 14 of Period 2 and Day 14 of Periods 3 and 4 to determine the Tmax.
Time Frame: up to 24 hours post morning dose on Days 1 and 14 of Period 2 and Day 14 of Periods 3 and 4
Population: No participants were enrolled in Part 2 of the study.
Arm/Group | MK-7145 10 mg (Part 2: Period 2) | MK-7145 16 mg | MK-7145 24 mg (Part 2: Period 4)
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Apparent Terminal Half-life (t1/2) of MK-7145 (Part 2)
Description: Blood samples taken at predose, 0.5, 1, 2, 5, 8, 12, 14 and 24 hours postdose on Days 1 and 14 of Period 2 and Day 14 of Periods 3 and 4 to determine the t1/2.
Time Frame: up to 24 hours post morning dose on Days 1 and 14 of Period 2 and Day 14 of Periods 3 and 4
Population: No participants were enrolled in Part 2 of the study.
Arm/Group | MK-7145 10 mg (Part 2: Period 2) | MK-7145 16 mg (Part 2: Period 3) | MK-7145 24 mg (Part 2: Period 4)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 33 days for each treatment period (Period 1includes a break of up to 25 days between Periods 1 and 2; Period 2 includes 14 days post last dose in Period 2). Post-trial period includes time from 14 days post last dose to last reported AE (~ 90 days)
Description: Population includes all participants who received at least one dose of the study drug. Adverse events (AEs) for the treatment period are reported by study drug taken during the active treatment periods. AEs for the post trial period are reported as one group. Part 1: Period 3 and Part 2: All periods were not conducted.
Groups:
- MK-7145 8 mg (Part 1:Period 1): Single daily dose of 8 mg MK-7145 for 5 days, capsules, orally administered in a fasted state
- Furosemide 40 mg (Part 1:Period 2): Two daily doses of one 40 mg Furosemide tablet for 5 days administered in a fasted state
- Post Trial: Participants who received at least one dose of study drug during Period 1 or 2 of Part 1 of the study
Arm/Group | MK-7145 8 mg (Part 1:Period 1) | Furosemide 40 mg (Part 1:Period 2) | Post Trial
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 1/11
Other Adverse Events (participants affected / at risk) | 10/11 | 5/10 | 3/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-7145 8 mg (Part 1:Period 1) (N=11) | Furosemide 40 mg (Part 1:Period 2) (N=10) | Post Trial (N=11)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-7145 8 mg (Part 1:Period 1) (N=11) | Furosemide 40 mg (Part 1:Period 2) (N=10) | Post Trial (N=11)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Application site inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Catheter site bruise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Catheter site swelling (General disorders) | 2 (2) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness postural (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Xeroderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (2) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study terminated early due to lack of efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.